CLINICAL TRIAL: NCT05320419
Title: The Effect of Amniotic Membrane Injection as An Addition to Physical Therapy in Patients With Rotator Cuff Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210711R
Record Dates: First submitted 2022-02-08; First posted 2022-04-11 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Tendinopathy; Ultrasonography
Keywords: Rotator cuff tear; rotator cuff tendinopathy; amniotic membrane; ultrasonography
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Injections; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotic membrane preparation and injection (AM group) (Active Comparator): The dehydrated AM product used in this study is derived from donated human placental tissue following healthy, live, caesarian section, full-term births which are then cleaned of blood under aseptic conditions. The product comes as a 20mg dry powder in a small vial stored at room temperature and mixed with 2 mL 0.9% sterile normal saline. Then the suspended AM will be injected to the injured tendon and the surrounding area with ultrasound-guidance via a 7cm, 23-gauge needle.
  Interventions: Other: Physiotherapy (PT group)
- Physiotherapy (PT group ) (Active Comparator): Physiotherapy includes hot pack, electric therapy and therapeutic exercise, which will be supervised by a senior physical therapist. The therapeutic exercise consists of active and passive stretching, and strengthening exercise of the rotator cuff, the shoulder girdle, and the pectoral muscles, and scapular stabilization exercise, 3 times a week, and will be continued for 12 weeks.
  Interventions: Other: Amniotic membrane preparation and injection (AM group)

INTERVENTIONS:
Other: Amniotic membrane preparation and injection (AM group) — The dehydrated AM product used in this study is derived from donated human placental tissue following healthy, live, caesarian section, full-term births which are then cleaned of blood under aseptic conditions. The product comes as a 20mg dry powder in a small vial stored at room temperature and mixed with 2 mL 0.9% sterile normal saline. Then the suspended AM will be injected to the injured tendon and the surrounding area with ultrasound-guidance via a 7cm, 23-gauge needle.
  Arms: Physiotherapy (PT group )
Other: Physiotherapy (PT group) — Physiotherapy includes hot pack, electric therapy and therapeutic exercise, which will be supervised by a senior physical therapist. The therapeutic exercise consists of active and passive stretching, and strengthening exercise of the rotator cuff, the shoulder girdle, and the pectoral muscles, and scapular stabilization exercise, 3 times a week, and will be continued for 12 weeks.
  Arms: Amniotic membrane preparation and injection (AM group)

SUMMARY:
Rotator cuff tear (RCT) is a commonly seen pathology in shoulder disease, which causes significant disability in daily living and work. Based on a cohort study of a large population, the prevalence of rotator cuff full-thickness tear was 20.7%. More broadly, the prevalence of rotator cuff abnormalities increased with age and up to 62% in population more than 80 years old. The pathophysiology of RCT could be attributed to extrinsic factors such as impingement by surrounding tissue and intrinsic factor such as tendon degeneration. According to previous study using histochemical and immunocytochemical techniques, fibrocartilaginous metaplasia, decreasing vascularity and fibroblast numbers were found in rotator cuff tear. Besides, the inflammatory response diminished as the tear size increased.

The treatment of RCT includes surgery and non-operative treatment. The prognosis depends on the symptoms, tear size, chronicity and other structures involvement. Previous meta-analysis study reported that the effectiveness between surgery and conservative treatment is similar in treating RCT. Therefore, relative rest, oral medication, physical therapy and injection therapy were commonly used in first-line treatments. When treating shoulder pain with injection therapy, steroid was often used at first for short-term pain relief and anti-inflammation. However, the potential cytotoxic effect was found and could be harmful in tendon repair. To accelerative the healing process of soft tissue injury, regenerative injection become more popular and expectable over past few years. A meta-analysis study reported the positive long-term effect of prolotherapy and platelet-rich plasma (PRP). More recently, bone marrow concentrate (BMC) and amniotic membrane (AM) have been used in soft tissue repair and many clinical studies are processing.

DETAILED DESCRIPTION:
Rotator cuff tear (RCT) is a commonly seen pathology in shoulder disease, which causes significant disability in daily living and work. Based on a cohort study of a large population, the prevalence of rotator cuff full-thickness tear was 20.7%. More broadly, the prevalence of rotator cuff abnormalities increased with age and up to 62% in population more than 80 years old. The pathophysiology of RCT could be attributed to extrinsic factors such as impingement by surrounding tissue and intrinsic factor such as tendon degeneration. According to previous study using histochemical and immunocytochemical techniques, fibrocartilaginous metaplasia, decreasing vascularity and fibroblast numbers were found in rotator cuff tear. Besides, the inflammatory response diminished as the tear size increased.

The treatment of RCT includes surgery and non-operative treatment. The prognosis depends on the symptoms, tear size, chronicity and other structures involvement. Previous meta-analysis study reported that the effectiveness between surgery and conservative treatment is similar in treating RCT. Therefore, relative rest, oral medication, physical therapy and injection therapy were commonly used in first-line treatments. When treating shoulder pain with injection therapy, steroid was often used at first for short-term pain relief and anti-inflammation. However, the potential cytotoxic effect was found and could be harmful in tendon repair. To accelerative the healing process of soft tissue injury, regenerative injection become more popular and expectable over past few years. A meta-analysis study reported the positive long-term effect of prolotherapy and platelet-rich plasma (PRP). More recently, bone marrow concentrate (BMC) and amniotic membrane (AM) have been used in soft tissue repair and many clinical studies are processing.

In recent decades, PRP was widely used in soft tissue regeneration. Though many studies had discussed the effect of PRP injections on pain and shoulder function in RCT, the effectiveness remains controversial. Some newer scaffolds including bovine collagen and amnio-derived membranes were also applied to the RCT in recent years. The AM was separated from a donor's placenta, and is a non-immunogenic structure. In previous animal study, amniotic epithelial cells could produce transforming growth factor-β (TGF-β), basic fibroblast growth factor (bFGF), epidermal growth factor (EGF), transforming growth factor-α (TGF-α), keratinocyte growth factor and hepatocyte growth factor. AM was found having anti-inflammatory, antimicrobial, antiviral effect, regulatory effect on angiogenesis and anti-scarring effcts. AM was revealed a pluripotent tissue which makes it potential in regenerative medicine. In some case series research, positive results was reported in pain and shoulder function in rotator cuff tears.

To the best of our knowledge, there has been limited evidence of regenerative injection by AM in treating patients with rotator cuff tear. The aim of this study is to evaluate the effect of single injection of AM in addition to physical therapy on pain and shoulder function.

ELIGIBILITY:
Inclusion Criteria:

1. . symptomatic rotator cuff tendinopathy, including partial-thickness tear or small (<1cm) full-thickness tear, proven by ultrasound
2. . duration of symptom longer than 1 month
3. . age ≥20 years old

Exclusion Criteria:

1. .fracture, dislocation, or arthritis of the shoulder
2. . previous shoulder joint surgery
3. . rotator cuff full-thickness tear with size ≥ 1cm
4. . calcification of rotator cuff tendons
5. . severe medical comorbidities, e.g., malignant neoplasms, blood dyscrasia, and serious infection, etc.
6. . pregnancy
7. . cognitive impairment (Mini-Mental Status Examination < 24).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale (VAS) | change between baseline and at 4 weeks, 12 weeks, and 24 weeks after the beginning of the treatment.
  The pain VAS during Neer test will be obtained using a horizontal line of 100 mm, with 0 on the left indicating no pain and 100 on the right indicating very severe pain. A pain VAS has been shown to be reliable and sensitive for quantifying pain, with test-retest reliability of >0.90.24 In previous studies of patients treated for various shoulder disorders, the responsiveness of VAS for pain was moderate to good.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | change between baseline and at 4 weeks, 12 weeks, and 24 weeks after the beginning of the treatment.
  The SPADI is a self-administered questionnaire to assess the pain and disability associated with shoulder diseases. It consists of 13 items being divided into 2 subclasses, 5 items for pain and 8 items for disabilities. The total SPADI score, which ranges between 0 and 100, is calculated by averaging the scores from the pain and disabilities subclasses. Good validity and reliability had been proved in previous studies.

OTHER OUTCOMES:
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) | change between baseline and at 4 weeks, 12 weeks, and 24 weeks after the beginning of the treatment.
  The ASES is a composite instrument, requiring both a physician assessment and a patient-completed portion; however, it is commonly presented as solely the patient-reported survey. This includes a section on pain (7 items) and a section on activities of daily living (10 items). Scores range from 0 to 100 with a higher score indicating a better shoulder condition. The minimal detectable change was 9.7 points, and the minimal clinically important difference was 6.4 points.
Range of motion. | change between baseline and at 12 weeks, and 24 weeks after the beginning of the treatment.
  The passive ROMs of the affected shoulder will be measured using a goniometer with the guidelines of the American Academy of Orthopedic Surgeons.22 This measurement includes abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 0 degrees of abduction. These ROM measurements of the shoulder using goniometer have been reported to have high inter-trial reliability when they are performed by the same physical therapist.
Ultrasound image of the rotator cuff of the affected shoulder | change between baseline and at 4 weeks, 12 weeks, and 24 weeks after the beginning of the treatment.
  EPIQ 5 (Phillips, USA) machine with a 18- to 4-MHz linear array transducer will be used for ultrasonographic examinations of the shoulder. The examination will be performed with the subjects in seated position and will be started from the biceps tendon, subscapularis tendon, supraspinatus tendon, infraspinatus tendon, and subacromial-subdeltoid bursa in both the transverse and longitudinal planes. AC joint will also be examined in the longitudinal plane.
Self-assessment of the treatment effect. | change between baseline and at 4 weeks, 12 weeks, and 24 weeks after the beginning of the treatment.
  Patient's evaluation of the treatment effect consists of the answer to one question: "Is the treatment effective?" scored on a Likert scale (very effective=5, effective=4, not effective=3, worse=2, much worse=1).

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan